CLINICAL TRIAL: NCT06295380
Title: Study of Motor Recovery and Biomechanical Adaptation Mechanisms in Amputee Patients Using an Immersive Virtual Reality System (CAREN)
Brief Title: Virtual Reality Rehabilitation to Promote Motor Recovery in Amputees
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Mirjam Bonanno, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CarenAmp
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Lower Limb Amputation Knee; Injuries; Biomechanical Lesion
Keywords: rehabilitation; virtual reality
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual environment practiced on the Caren (Experimental): Caren virtual training phase plus conventional physiotherapy phase
  Interventions: Behavioral: Virtual environment practiced on the Caren
- Conventional physiotherapy (Active Comparator): Conventional physiotherapy phase plus Caren virtual training phase
  Interventions: Behavioral: Conventional physiotherapy

INTERVENTIONS:
Behavioral: Virtual environment practiced on the Caren — The virtual environment practised on the Caren will make the scenario totally immersive and allow the subject to perform the motor task by recruiting muscles according to a motor coordination scheme different from the traditional one.
  Arms: Virtual environment practiced on the Caren
Behavioral: Conventional physiotherapy — Conventional physiotherapy
  Arms: Conventional physiotherapy

SUMMARY:
Interventional, non-pharmacological crossover study aimed at identify statistically significant differences in postural stability and spatio-temporal gait cycle parameters in patients with lower limb amputation by means of taskoriented rehabilitation training and multisensory feedback generated by an immersive RV environment, aiming at the enhancement of use-dependent brain plasticity. These changes will be compared between the two groups examined, respectively experimental (Caren virtual training phase plus conventional physiotherapy phase) and control (conventional physiotherapy phase plus Caren virtual training phase).

DETAILED DESCRIPTION:
Primary objectives: Evaluation of biomechanical and spatio-temporal asymmetries in gait in subjects with lower limb amputation by motion capture systems; improvement of postural stability and gait cycle in patients with lower limb amputation by "task-oriented" rehabilitation training and multisensory feedback generated by an immersive virtual reality environment, aiming at the enhancement of use-dependent brain plasticity; improving body weight distribution on both lower limbs, during static and dynamic activities, through more effective control of the body's centre of gravity. Secondary objectives include improving mood, psycho-social wellbeing and quality of life in lower limb amputees.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower limb amputation
* ability to walk independently
* age between 18 and 75 years
* absence of severe comorbidities that may interfere with treatment

Exclusion Criteria:

* presence of severe neurological and psychiatric disorders
* walking with aids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Kinematic data | seven months
  From the gait analysis, the investigators will obtain kinematic data, including spatial and temporal parameters measured during standing acquisition and kinematic analysis evaluated from the walking trials recordings.
Kinetic data | seven months
  From the gait analysis, the investigators will obtain kinetic data concerning the joint moments and powers, joints moments and powers normalized by the subject's weight (Newton*meter/kg e Watt/kg) and ground reaction forces reported in percentage to the body weight will be averaged across all cycles for each subject for each evaluating session.
Electromyography | seven months
  From the gait analysis, the investigators will obtain electromyographic data on electromyopgraphic signals, regarding muscle contraction, which will be recorded with surface electrodes. The raw signals (millivolts) will be filtered with a band pass filter (20 - 450 Hz) and time-normalized for the duration of the gait cycle (% gait cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Paladina, PT, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No
After the data collection we will report anonymised data on public repository